CLINICAL TRIAL: NCT06246162
Title: Mitoxantrone Hydrochloride Liposome Combination Regimen in the Treatment of High-risk/Extramedullary Multiple Myeloma:A Single-arm, Single-center, Prospective Clinical Trial
Brief Title: Mitoxantrone Hydrochloride Liposome Combination Regimen in the Treatment of High-risk/Extramedullary Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Hongming Huang, professor, Affiliated Hospital of Nantong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-TDFY-052
Record Dates: First submitted 2023-11-14; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipo-MIT combination regimen group (Experimental): Initial diagnosis induction treatment regimen Lipo-MIT +VD (VMD):
  Mitoxantrone Hydrochloride Liposome: 10 mg, d1, d15, intravenous infusion; Bortezomib: 1.3mg/m2 d1, 4, 8, 11, subcutaneous injection; Dexamethasone: 20 mg/d, orally on days 1, 2, 4, 5, 8, 9, 11, and 12. Every 4 weeks constitutes a cycle, and 4 cycles of VMD regimen induction therapy are performed.
  Reinduction therapy regimen after relapse Lipo-MIT + PD (PMD):
  Mitoxantrone Hydrochloride Liposome: 10 mg, d1, d15, intravenous infusion; Pomalidomide: 4 mg/d d1-d21, orally; Dexamethasone: 20 mg/d, orally on days 1, 2, 4, 5, 8, 9, 11, and 12. Every 4 weeks constitutes a cycle, and 4 cycles of PMD regimen induction therapy are performed.
  Interventions: Drug: Lipo-MIT combination regimen

INTERVENTIONS:
Drug: Lipo-MIT combination regimen — Initial diagnosis induction treatment regimen Lipo-MIT +VD (VMD):
  Mitoxantrone Hydrochloride Liposome: 10 mg, d1, d15, intravenous infusion; Bortezomib: 1.3mg/m2 d1, 4, 8, 11, subcutaneous injection; Dexamethasone: 20 mg/d, orally on days 1, 2, 4, 5, 8, 9, 11, and 12. Every 4 weeks constitutes a cycle, and 4 cycles of VMD regimen induction therapy are performed.
  Reinduction therapy regimen after relapse Lipo-MIT + PD (PMD):
  Mitoxantrone Hydrochloride Liposome: 10 mg, d1, d15, intravenous infusion; Pomalidomide: 4 mg/d d1-d21, orally; Dexamethasone: 20 mg/d, orally on days 1, 2, 4, 5, 8, 9, 11, and 12. Every 4 weeks constitutes a cycle, and 4 cycles of PMD regimen induction therapy are performed.

SUMMARY:
To evaluate the efficacy and safety of mitoxantrone Hydrochloride Hydrochloride Liposome combination regimen in the treatment of high-risk/extramedullary multiple myeloma

DETAILED DESCRIPTION:
This study is expected to be carried out from November 2023 to November 2026. About 30 patients with high-risk/extramedullary multiple myeloma will receive mitoxantrone Hydrochloride Liposome combination regimen treatment. After evaluating of efficacy and safety of treatment, the principal investigator will write and publish the paper.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed with high-risk multiple myeloma (del17p, t (4; 14), t (14; 16), 1q21 by FISH test) or extramedullary multiple myeloma; 2. Age: 18-70 years old (including 18 and 70 years old), regardless of gender; 3. Eastern Cooperative Oncology Group physical performance score (ECOG): 0-2 points; 4. Expected survival ≥3 months; 5. Have "measurable lesions": extramedullary lesions ≧1.0cm or more; serum M protein ≥10g/L and/or 24-hour urine M protein ≥200mg; 6. Blood routine: neutrophil count ≥1.0×109/L; for patients with plasma cells in bone marrow >50%, 0.5×109/L≤neutrophil count <1.0×109/L is allowed. For patients with platelets ≥100×109/L; plasma cells in bone marrow >50%, 50×109/L≤platelets <100×109/L; hemoglobin >8g/dL; 7. Liver function: AST and ALT ≤ 2.5 times the upper limit of normal value (for the same age group), or ≤ 5 times the upper limit of normal value in the presence of liver metastasis; total bilirubin ≤ 1.5 times the upper limit of normal value; creatinine ≤ 2.5 mg/dL ; 8. Patients receiving localized radiation therapy, with or without concomitant steroids, for pain control or spinal cord/nerve root compression treatment are eligible. More than 4 weeks since the last radiotherapy treatment; 9. Sign the informed consent form.

Exclusion Criteria:

* 1. Impaired heart function or suffering from significant heart disease, including but not limited to:

  1. Myocardial infarction or viral myocarditis occurred within 6 months before screening;
  2. There are heart diseases that require treatment at the time of screening, such as unstable angina, chronic congestive heart failure (NYHA ≥ grade 2), arrhythmia, valvular disease, etc. or persistent cardiomyopathy;
  3. QTc interval >480ms or suffering from long QTc syndrome during screening;
  4. The cardiac ejection fraction is lower than 50% or lower than the lower limit of the examination value range of the research center during screening.

     2. Active infection of hepatitis B and hepatitis C (hepatitis B virus surface antigen is positive and hepatitis B virus DNA exceeds 1x103 copies/mL; hepatitis C virus RNA exceeds 1x103 copies/mL); 3. Human immunodeficiency virus (HIV) infection (HIV antibody positive); 4. Suffer from uncontrollable bacterial infection, fungal infection or viral infection that requires systemic treatment within 1 week before the administration of the study drug; 5. Women who are pregnant or breastfeeding; 6. Peripheral neuropathy or pain of grade 2 (CTCAE5.0) or above before treatment; 7. Received systemic chemotherapy within 28 days before the first dose; 8. Relapsed patients are resistant to pomalidomide in previous treatment or cannot accept pomalidomide treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  objective remission rate

SECONDARY OUTCOMES:
2-years PFS | 2 years
  2-years progression-free survival rate
2-years OS | 2 years
  2-years overall survival rate
2-years extramedullary relapse rate | 2 years
  2-years extramedullary relapse rate
DoR | 2 years
  duration of response
TTNT | 2 year
  time to the next treatment
MRD negative conversion rate | 6 months
  minimal residual disease negative conversion rate

CONTACTS AND LOCATIONS:
Overall Officials: Hongming Huang, PhD, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Not planning sharing at present